CLINICAL TRIAL: NCT01287052
Title: Nitrous Oxide for Acute Pediatric Migraine Pain Management in the Emergency Room
Brief Title: Nitrous Oxide for Acute Migraine Pain in the Emergency Room (ED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1101-006
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2014-04

CONDITIONS: Migraine; Pain
Keywords: Migraine; Pediatric; Adolescent; Nitrous Oxide
MeSH Terms: conditions — Migraine Disorders; Pain | interventions — Nitrous Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitrous Oxide (Experimental)
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous Oxide — Once consent is obtained, the research assistant will notify the charge RN and MD of the patient's study participation. The patient will then be placed in a treatment room and nitrous oxide will be administered per the existing protocol. Each participant will be given nitrous oxide until he/she reports a pain score of zero or up to fifteen minutes. Study subjects will be asked to rate their pain on a scale of 0-10 before the treatment and after the treatment, the time duration of administering nitrous oxide will be recorded. In addition, the pain scores at 30, 60, 90, and 120 minutes post baseline measurement will be collected in order to evaluate the sustained effect of nitrous oxide in treating acute migraine pain. Someone from the study will also make a follow-up phone call 24 - 48 hours to see if pain relief persisted.

SUMMARY:
BACKGROUND Migraine headaches account for 8-18% of all headaches seen in pediatric emergency rooms. Standard treatment includes IV pain medications, anti-emetics, and IV fluids. Nitrous oxide has analgesic properties similar to those of opioids and is easy to administer. It has been shown in two small studies to be effective in treating migraine headaches.

RESEARCH QUESTION Does nitrous oxide act as a safe, less invasive, and effective treatment of acute migraine headaches in children and adolescents presenting to an Emergency Department?

DESIGN This is a prospective non-randomized self-controlled study. Repeated measures will be taken to examine change in pain scores before and after nitrous oxide treatment.

METHODS Each participant will be given nitrous oxide until he/she reports a pain score of zero or up to fifteen minutes. Study subjects will be asked to rate their pain on a scale of 0-10 before the treatment and after the treatment at multiple time-points.

ELIGIBILITY:
Inclusion Criteria:

* During the study enrollment period, eligible subjects will be English-speaking children and adolescents
* Between the ages of 8 - 18 years (inclusive)
* With history of migraine present for at least one year
* With previous migraine headaches conforming to ICHD-II diagnostic criteria
* Able to give assent according to institutional guidelines, and
* Have parental consent to participate.

Exclusion Criteria:

* Any patients will be excluded if he/she
* Has had any neurosurgical interventions
* Has underlying seizure disorders
* Presents with a headache of a different quality than their other migraines
* Has contraindications to nitrous oxide
* Unable to complete the pain assessment
* Does not have a dependable contact number for the follow-up call

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Decrease in the acute migraine pain in children and adolescents presenting to an Emergency Department | within 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Hoogerland, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota, United States